CLINICAL TRIAL: NCT04075383
Title: Immediate and Immediate-delayed Implants in the Esthetic Area: 12-months Randomized Controlled Trial
Brief Title: Immediate and Early Single Dental Implants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11851319.9.0000.5347
Record Dates: First submitted 2019-06-27; First posted 2019-08-30 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Single Tooth Lost; Dental Implant
Keywords: dental implant; esthetics; quality of life
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: randomised controlled parallel clinical trial
Who Masked: Outcomes Assessor
Masking Description: Researchers involved in the assessment of all outcomes will be not aware of the randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate dental implant (Other): The implant is installed immediately after tooth extraction.
  Interventions: Procedure: immediate dental implant
- immediate-delayed dental implant (Other): The implant is installed 8 weeks after tooth extraction.
  Interventions: Procedure: immediate-delayed dental implant

INTERVENTIONS:
Procedure: immediate dental implant — Replacement of a lost tooth with a titanium screw retained in the alveolar bone in the same session of tooth extraction.
  Arms: immediate dental implant
Procedure: immediate-delayed dental implant — Replacement of a lost tooth with a titanium screw retained in the alveolar bone 8 weeks after tooth extraction.
  Arms: immediate-delayed dental implant

SUMMARY:
The objective of the research project will be to compare immediate and early unitary implants for the rehabilitation of missing teeth in the upper aesthetic region. A randomized controlled trial will be conducted in parallel with 120 individuals (60 per group) who are above 18 years of age, periodontally healthy, and who need to perform only one unit implant in the upper aesthetic region between the second premolars. In the immediate implant group, the tooth will be extracted in a minimally traumatic manner and the implant will be installed immediately after the fresh alveolus. Bovine bone replacement will be inserted into the gap between implant and vestibular wall of the alveolus, and an immediate temporary will be installed immediately. The provisional will be maintained for 3 months when the definitive crown will be made. In the early implant group, the tooth will be extracted, and after 2 months the implant will be installed with the use of bovine bone substitute to restore the buccal bone contour. The implant will be submerged, and 3 months of osseointegration will be performed reopening and final crown making. In both groups, the individuals will be followed for 1 year after the installation of the definitive crown. The outcomes evaluated will be patient satisfaction (main outcome), gingival phenotype, visible plaque, depth of probing, submucosal bleeding, proximal radiographic bone level, tomographic vestibular bone volume, perimplant clinical aesthetic indexes (Esthetic Pink Score and Papillary Index), evaluation three-dimensional tissue from intra-oral scanning and 3D printing, implant-related quality of life, and early and late implantation failures. Linear and logistic models of generalized estimating equations that take into account the longitudinal character of the study will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old who require only one single implant in the upper aesthetic area between the second premolars will be included.
* The region from which the tooth will be extracted should have bone quality and quantity compatible with implant placement with a minimum diameter and length of 3.0 mm and 8.0 mm, respectively.

Exclusion Criteria:

* Who present compromise immunology of any nature;
* Who have been exposed to head and neck radiotherapy;
* Who have uncontrolled diabetes (glycated hemoglobin above 6.5 mg/dL);
* Who present active periodontitis, defined by the presence of bleeding on probing >10% and probing depth and clinical attachment loss > 4mm;
* Who have performed or are being treated with intravenous bisphosphonates.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-22 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction: questionnaire | Up to 24 months
  satisfaction with treatments by questionnaire in a VAS scale
tridimensional tissue changes | Up to 24 months
  3D measurements obtained in oral scanning
Buccal bone level | Up to 24 months
  CBCT analysis of the buccal bone

SECONDARY OUTCOMES:
Pink esthetic score | Up to 24 months
  Evaluation of the clinical esthetic outcome of soft tissues in 7 parameters recorded from 0 to 2, summing up a total of 14 points
White esthetic score | Up to 24 months
  Evaluation of the clinical esthetic outcome of prosthetic crowns recorded from 0 to 2, summing up a total of 14 points
Implant failure | Up to 24 months
  Failure defined as loss of implant
Oral health related quality of life: OHIP-14 | Up to 24 months
  Questionnaire assessing 14 questions of quality of life in a likert scale summing up a total of 48 points
dental plaque | Up to 24 months
  Plaque accumulation at the crowns
Pocket depth | Up to 24 months
  Measured in millimetres
Bleeding | Up to 24 months
  Bleeding after probing

CONTACTS AND LOCATIONS:
Overall Officials: Alex Haas, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Alex Haas, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No